CLINICAL TRIAL: NCT01308879
Title: Effects of Routine Feedback to Clinicians on Youth Mental Health Outcomes: A Randomized Cluster Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Leon Lowenstein Foundation Inc. (Other)
Responsible Party: Leonard Bickman, Principal Investigator, Center for Evaluation and Program Improvement, Peabody College, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 070342; R01MH068589 (NIH)
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Mental Health Wellness 1; Psychosocial Problem
Keywords: Contextualized Feedback System (CFS); Mental health outcomes; Quality improvement; Feedback; Clinical trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weekly feedback (Experimental): After clinical questionnaires are entered into the system (CFStm), an automated online report is available weekly to clinicians in the experimental group that shows current mental health status of youths, alerts, and trends over time based on youth, caregiver, and clinician responses. Reports also show some clinical data on caregivers.
  Interventions: Behavioral: Contextualized Feedback Systems (CFS)tm
- No feedback (Other): Clinicians in the control group do not have access to weekly feedback. Instead, they receive reports every 90 days after the youth is enrolled in CFStm. Because the average duration of CFS enrollment was 3.8 months, many youths would have been discharged before the first 90-day report became available three months after treatment start. Thus, we considered the 90-day feedback group to be essentially a no-feedback group.
  Interventions: Behavioral: Contextualized Feedback Systems (CFS)tm

INTERVENTIONS:
Behavioral: Contextualized Feedback Systems (CFS)tm — After clinical questionnaires are entered, an automated feedback report is available online weekly to clinicians (and supervisors) in the experimental group. The report shows current mental health status of youths, alerts, and trends over time. Reports also show some clinical data on youths' caregivers.

SUMMARY:
The purpose of this clinical trial was to test the hypothesis that clients of clinicians who were scheduled to receive weekly feedback on their clients' progress would improve faster than clients of clinicians who were not scheduled to receive weekly feedback.

DETAILED DESCRIPTION:
The primary approach to improving psychosocial treatment for youths has been to implement evidence-supported treatments (ESTs) in community services. However, this approach has not produced clear cut results of effectiveness. A recently developed alternative is to improve outcomes through routine measurement and feedback to clinicians and supervisors. The investigators used a cluster randomized experiment with 28 sites affiliated with a national behavioral health organization to assess whether clients of clinicians who were scheduled to receive weekly feedback on their clients' progress would improve faster than clients of clinicians who were not scheduled to receive weekly feedback.

ELIGIBILITY:
Inclusion Criteria:

* all youths 11-18 years old, entering treatment as usual, home-based services through the service provider. Youths' primary caregiver and clinician also participate.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 356 (Actual)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Symptoms and Functioning Severity Scale | The SFSS is completed at intake by youths and caregivers, then by youths, caregivers, and clinicians at the 1st treatment session and every other session (week) thereafter for as long as the youth is enrolled in the intervention (CFS).
  The SFSS is part of a battery of clinical measures (Peabody Treatment Progress Battery:PTPB) developed by the researchers. It assesses change in closely-timed repeated measurements. Parallel forms are completed by youths, caregivers, and clinicians at the end of treatment sessions. The SFSS includes 32 items that ask the respondent to rate how frequently in the last two weeks the youth experienced emotions or exhibited behaviors linked to typical mental health disorders for youths (e.g., ADHD, conduct disorder, depression).

SECONDARY OUTCOMES:
Brief Multidimensional Students' Life Satisfaction Scale-CEPI (BMSLSS-CEPI) | The BMSLSS-CEPI is completed by the youth at intake, at the 2nd treatment session, and every 8 weeks thereafter for as long as the youth is enrolled in the intervention (CFS).
  The BMSLSS-CEPI is a revised version of the Brief Multidimensional Students' Life Satisfaction Scale (Seligson, Huebner, & Valois, 2003). The BMSLSS-CEPI was designed to assess global life satisfaction as well as domain specific satisfaction with family, friends, school, self and living environment. Life satisfaction may be targeted directly or indirectly with treatment and thus can be thought of as a positive, or strengths-based, indicator of treatment progress (outcome).
The Children's Hope Scale (CHS) | The CHS is completed by the youth at intake and every 8 weeks thereafter for as long as the youth is enrolled in the intervention (CFS).
  The CHS (Snyder et al., 1997), a public domain measure used with youth in this study, assesses youth hopefulness. The measure asks youths to report on their ability to generate paths toward goals and persevere toward those goals. Youth hopefulness is conceptually an important factor in the successful treatment of emotional or behavioral disorders, constituting an outcome that may be affected by the treatment process.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Bickman, Ph.D., Principal Investigator — Center for Evaluation and Program Improvement, Vanderbilt University
Locations (1):
- 28 sites in 10 states affiliated with Providence Service Corporation (location info is for corporate office), Tucson, Arizona, United States